CLINICAL TRIAL: NCT05498025
Title: The Effect of a Charcoal Deactivation Pouch on Opioid Disposal After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Michael J. Paglia, MD PhD, Principal Investigator, Geisinger Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0487
Record Dates: First submitted 2022-03-31; First posted 2022-08-11 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Pain, Acute; Opioid Misuse; Obstetric Pain; Cesarean Section Complications
Keywords: opioid disposal; drug deactivation; Deterra
MeSH Terms: conditions — Acute Pain; Opioid-Related Disorders; Labor Pain

STUDY DESIGN:
Intervention Model Description: This is a prospective single arm interventional pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Activated charcoal pouch (Experimental): The patients in this arm will receive an activated charcoal pouch (Deterra Medium Pouch, UPC #: 850006727001, Verde Environmental Technologies, Minnetonka, MN) for disposal of their opioids after their cesarean delivery pain has resolved.
  Interventions: Other: Deterra activated charcoal pouch

INTERVENTIONS:
Other: Deterra activated charcoal pouch — drug disposal pouch

SUMMARY:
Background: There is scarce literature investigating how patients dispose of unused opioid supplies after their cesarean postoperative pain has faded. The Office of the Surgeon General has identified research on the prevention of opioid use disorder area as well as research on the management of pain as a "Surgeon General Priority" that needs urgent investigation.

Hypothesis: At least 33% of postpartum women discharged home with an opioid prescription and a drug deactivation pouch will use the pouch to dispose of remaining opioids within 30 days of delivery.

Methods: This is a prospective single arm interventional pilot study.

ELIGIBILITY:
Inclusion criteria:

* Age 18+ at time of enrollment, per ERM
* Delivered ≥26.0 weeks, per ERM
* Status post low transverse cesarean delivery, per ERM
* Physically located on labor & delivery and is postpartum day #1 or #2 at time of enrollment, per ERM
* Opioid prescription has been sent (per ERM) or will be sent (per obstetric team).

Exclusion criteria:

* Positive urine toxicology anytime in pregnancy for non-prescription opioids, fentanyl, amphetamines, benzodiazepines, cannabinoids, LSD, or cocaine, per ERM.
* Buprenorphine or methadone Rx, per ERM
* Patient preferred communication language not English, per ERM
* Documented history, per ERM:

  * Cannabinoid use disorder
  * Hypnotic use disorder
  * Opioid use disorder
  * Stimulant use disorder
  * Fibromyalgia
  * Sickle cell anemia
  * Lumbar disc herniation
  * Multiple sclerosis
  * Trigeminal neuralgia
  * Active cancer
  * Complex regional pain syndrome
  * Systemic lupus erythematosus
  * Rheumatoid arthritis

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
Actual pouch use | 30 days
  The percentage of women who used the pouch to dispose of opioids in the home 30 days after delivery (%)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Paglia, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No